CLINICAL TRIAL: NCT06406998
Title: Maternal and Offspring Outcomes in Pregnant Women With Pre-existing Atherosclerotic Cardiovascular Disease: A Nationwide Mother-Child Cohort Study
Brief Title: Maternal and Offspring Outcomes in Pregnant Women With Pre-existing ASCVD
Acronym: CVD_OBS
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ki Hong Choi, Associate Professor, Samsung Medical Center
Other Study IDs: CVD_OBS
Record Dates: First submitted 2024-05-04; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Pregnancy Complications; Adverse Cardiac Event; Adverse Birth Outcomes
Keywords: Atherosclerotic cardiovascular disease; Major adverse cardiac and cerebrovascular event; Adverse pregnancy outcome; Adverse birth outcomes
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women with pre-existing atherosclerotic cardiovascular disease: Among the total cohort, pregnant women with pre-existing atherosclerotic cardiovascular disease were selected (N=145,315).
  Interventions: Other: Pre-existing atherosclerotic cardiovascular disease
- Matched cohort: Among the total cohort, 1:4 matched offspring born to women without pre-existent atherosclerotic cardiovascular disease using a propensity score were generated (N=581,260).

INTERVENTIONS:
Other: Pre-existing atherosclerotic cardiovascular disease — Presence of pre-existing atherosclerotic cardiovascular disease
  Groups: Pregnant women with pre-existing atherosclerotic cardiovascular disease

SUMMARY:
A growing body of evidence supports associations between cardiovascular health and adverse pregnancy outcome and between adverse pregnancy outcome and atherosclerotic cardiovascular disease and builds on the well-established pathways known to exist between cardiovascular health and atherosclerotic cardiovascular disease across the life course and intergenerationally. Furthermore, previous studies frequently lack comprehensive long-term follow-up, making it difficult to assess the enduring impacts of maternal cardiovascular health on postpartum outcomes and long-term maternal and child health.

DETAILED DESCRIPTION:
the current study aimed to evaluate the associations between maternal pre-existent atherosclerotic cardiovascular disease and adverse pregnancy outcomes, and the combined effect of maternal pre-existent atherosclerotic cardiovascular disease and adverse pregnancy outcomes on the risk of long-term adverse events of offspring.

ELIGIBILITY:
Inclusion Criteria:

* Women with live birth from Korea (between January 1, 2005 to December 31, 2019)

Exclusion Criteria:

* None

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: All womens with live birth from Korea
Sampling Method: Non-Probability Sample
Enrollment: 5461222 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurence of post-partum MACCE | up to 5 years
  major adverse cardiac and cerebrovascular event

SECONDARY OUTCOMES:
Occurence of All-cause death | up to 5 years
  Death from any causes
Occurence of myocardial infarction | up to 5 years
  Myocarrdial infarction
Occurence of revascularization | up to 5 years
  percutaneous coronary intervention or coronary artery bypass grafting
Occurence of stroke | up to 5 years
  Ischemic or hemorrhagic stroke
Occurence of adverse pregnancy outcome | At delivery
  preterm delivery, pre-eclampsia or eclampsia, other hypertensive disorder of pregnancy, small-for-gestational-age, and gestational diabetes
Occurence of major congenital malformation in offspring | At delivery
  congenital malformation in offspring
Occurence of neonatal adverse events in offspring | within 30 days
  transient tachypnea, respiratory distress syndrome, necrotizing enterocolitis, intraventricular hemorrhage, bronchopulmonary dysplasia, and sepsis
Occurence of adverse infant events in offspring | Within 1 year
  admission to intensive care unit and occurrence of seizure events
Occurence of neurodevelopmental disorders | up to 5 years
  autism spectrum disorder, attention-deficit/hyperactivity syndrome, cerebral palsy, any developmental delay including motor or cognitive delay, epileptic and febrile seizures and tics, and stereotypic behavior

CONTACTS AND LOCATIONS:
Overall Officials: Ki Hong Choi, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kang D, Heo J, Choi KH, Park T, Sung JH, Park TK, Lee JM, Cho J, Yang JH, Song YB, Hahn JY, Choi SH, Gwon HC, Oh SY. Association of maternal pre-existing atherosclerotic cardiovascular disease and neonatal and long-term offspring outcomes: a nationwide mother-child paired cohort. Hum Reprod Open. 2025 Nov 25;2025(4):hoaf074. doi: 10.1093/hropen/hoaf074. eCollection 2025. PMID 41383953